CLINICAL TRIAL: NCT03338439
Title: Glyco-metabolic Control, Inflammation Markers and Cardiovascular Outcomes in Diabetic Patients on Insulin Pump or Multiple Daily Injection
Brief Title: Insulin Pump vs Multiple Daily Injection on Cardiovascular Outcomes (ITALICO)
Acronym: ITALICO
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, Clinical Professor, University of Pavia
Other Study IDs: 20170003557
Record Dates: First submitted 2017-11-02; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CSII: CSII: patients with continuous subcutaneous insulin infusion
  Interventions: Device: CSII
- MDI: MDI: patients with multi-daily injections

INTERVENTIONS:
Device: CSII — This retrospective, observational trial will evaluate 104 diabetic patients with prior treatment with MDI initiating CSII therapy compared to 109 diabetic patients continuing MDI.
  Groups: CSII

SUMMARY:
The aim of this study was to evaluate if the positive effects recorded on glycemic control with CSII were maintained on the long term compared to multi-daily injections (MDI). The secondary objective was to evaluate if there is a reduction of type and number of cardiovascular events (CV) in CSII group compared to MDI group after 8 years of observation. This retrospective, observational trial evaluated 104 diabetic patients with prior treatment with MDI initiating CSII therapy compared to 109 diabetic patients continuing MDI.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 1 or 2 diabetes with prior treatment with MDI initiating CSII therapy with tubed insulin pumps
* patients type 1 or 2 diabetes with prior treatment with MDI continuing MDI
* patients attending the center for at least 8 years

Exclusion Criteria:

* patients not taking insulin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 and type 2 diabetes mellitus taking insulin
Sampling Method: Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Fasting glycemia | Change from Baseline, at 4 years and at 8 years
  Carbohydrate metabolism
Postprandial glycemia | Change from Baseline, at 4 years and at 8 years
  Carbohydrate metabolism
Glycated haemoglobin | Change from Baseline, at 4 years and at 8 years
  Index of glycemic compensation
Total Cholesterol | Change from Baseline, at 4 years and at 8 years
  Lipid metabolism
HDL-Cholesterol | Change from Baseline, at 4 years and at 8 years
  Lipid metabolism
Triglycerides | Change from Baseline, at 4 years and at 8 years
  Lipid metabolism
LDL-Cholesterol | Change from Baseline, at 4 years and at 8 years
  Lipid metabolism
Systolic Blood Pressure | Change from Baseline, at 4 years and at 8 years
  Haemodynamic parameter
Diastolic Blood Pressure | Change from Baseline, at 4 years and at 8 years
  Haemodynamic parameter

SECONDARY OUTCOMES:
Cardiovascular event | Change from Baseline, at 4 years and at 8 years
  Atrial fibrillation
Cardiovascular event | Change from Baseline, at 4 years and at 8 years
  Premature Ventricular Contractions
Cardiovascular event | Change from Baseline, at 4 years and at 8 years
  Acute Coronary Infarction
Cardiovascular event | Change from Baseline, at 4 years and at 8 years
  Angina Pectoris
Cardiovascular event | Change from Baseline, at 4 years and at 8 years
  Pericarditis
Cerebrovascular event | Change from Baseline, at 4 years and at 8 years
  Ischemic Stroke
Vascular event | Change from Baseline, at 4 years and at 8 years
  Peripheral Vascular Ischemia

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Matteo Foundation, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: No